CLINICAL TRIAL: NCT02054520
Title: A Phase 2b Study of Immune Checkpoint Inhibition With or Without Dorgenmeltucel-L (HyperAcute Melanoma) Immunotherapy for Stage IV Melanoma Patients
Brief Title: Immunotherapy Study for Patients With Stage IV Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Withdrawal of IND
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NLG0304; 1303-1217 (Other: Office of Biotechnology Activities (OBA))
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Results first posted 2020-04-29 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-03

CONDITIONS: Stage IV Melanoma; Metastatic Melanoma
Keywords: Stage IV; metastatic melanoma
MeSH Terms: conditions — Melanoma | interventions — ATF7IP protein, human; Immunotherapy; Ipilimumab; pembrolizumab; Nivolumab

ARMS (6):
- Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab (Experimental): Arm 1A will receive ipilimumab at 3 mg/kg given every 3 weeks for 4 weeks and 300 Million HyperAcute®-Melanoma (HAM) Immunotherapy cells per each immunization, given every week for 4 weeks, every 2 weeks for 5 months, every month for 6 months, and every 3 months for one year.
  Interventions: Drug: HyperAcute®-Melanoma (HAM) Immunotherapy; Drug: Ipilimumab
- Arm 2A Ipilimumab Alone (Active Comparator): Arm 2A will receive ipilimumab alone at 3 mg/kg every 3 weeks for a total of four doses.
  Interventions: Drug: Ipilimumab
- Arm 1B HyperAcute®-Melanoma (HAM) + nivolumab (Experimental): Arm 1B will receive nivolumab alone at 3 mg/kg given every 2 weeks and 300 Million HyperAcute®-Melanoma (HAM) Immunotherapy cells per each immunization, given every week for 4 weeks, every 2 weeks for 5 months, every month for 6 months, and every 3 months for one year.
  Interventions: Drug: HyperAcute®-Melanoma (HAM) Immunotherapy; Drug: Nivolumab
- Arm 2B Nivolumab alone (Active Comparator): Arm 2B will receive nivolumab alone at 3 mg/kg given every 2 weeks
  Interventions: Drug: Nivolumab
- Arm 1C HyperAcute®-Melanoma (HAM) + pembrolizumab (Experimental): Arm 1C will receive pembrolizumab at 2 mg/kg given every 3 weeks and 300 Million HyperAcute®-Melanoma (HAM) Immunotherapy cells per each immunization, given every week for 4 weeks, every 2 weeks for 5 months, every month for 6 months, and every 3 months for one year.
  Interventions: Drug: HyperAcute®-Melanoma (HAM) Immunotherapy; Drug: Pembrolizumab
- Arm 2C Pembrolizumab alone (Active Comparator): Arm 2C will receive pembrolizumab at 2 mg/kg given every 3 weeks
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: HyperAcute®-Melanoma (HAM) Immunotherapy
  Other Names: HyperAcute®-Melanoma; HAM; Dorgenmeltucel-L
  Arms: Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab; Arm 1B HyperAcute®-Melanoma (HAM) + nivolumab; Arm 1C HyperAcute®-Melanoma (HAM) + pembrolizumab
Drug: Ipilimumab
  Other Names: YERVOY; MDX-010; MDX-101
  Arms: Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab; Arm 2A Ipilimumab Alone
Drug: Pembrolizumab
  Other Names: Keytruda
  Arms: Arm 1C HyperAcute®-Melanoma (HAM) + pembrolizumab; Arm 2C Pembrolizumab alone
Drug: Nivolumab
  Other Names: Opdivo
  Arms: Arm 1B HyperAcute®-Melanoma (HAM) + nivolumab; Arm 2B Nivolumab alone

SUMMARY:
The purpose of this study is to examine the effectiveness of immune checkpoint inhibitors (drugs called ipilimumab, nivolumab, or pembrolizumab), either given alone, or in combination with the experimental immunotherapy drug, dorgenmeltucel-L, for melanoma. We hypothesize that this form of combinatorial immunotherapy will result in tumor stabilization or shrinkage, significant prolongation of progression-free, disease-free or overall survival compared to the use of immune checkpoint inhibitors alone.

DETAILED DESCRIPTION:
According to statistics of the American Cancer Society, an estimated 73,800 individuals will be diagnosed with melanoma and 9,900 will die of the disease in 2015 in the Unites States despite current therapy. This protocol attempts to exploit an approach to melanoma immunotherapy using a naturally occurring barrier to xenotransplantation in humans to increase the effectiveness of immunizing patients against their melanoma. The expression of the murine (1,3)galactosyltransferase [alpha(1,3)GT] gene results in the cell surface expression of (1,3)galactosyl-epitopes (alpha-gal) on membrane glycoproteins and glycolipids. These epitopes are the major target of the hyperacute rejection response that occurs when organs are transplanted from non-primate donor species into man. Human hosts often have pre-existing anti-alpha-gal antibodies that bind alpha-gal epitopes and lead to rapid activation of complement and cell lysis. The pre-existing anti-alpha-gal antibodies found in most individuals are thought to be due to exposure to alpha-gal epitopes that are naturally expressed on normal gut flora leading to chronic immunological stimulation.

These antibodies may comprise up to 1% of serum IgG. In this phase 2b study, patients with advanced stage melanoma will receive immune checkpoint inhibition consisting of ipilimumab, nivolumab, or pembrolizumab per the treating physician's standard of care. In addition to the immune checkpoint therapy, half of the patients will also receive dorgenmeltucel-L. Dorgenmeltucel-L is composed of irradiated allogeneic melanoma cell lines (HAM-1, HAM-2 and HAM-3). These cell lines have been transduced with a recombinant Moloney murine leukemia virus (MoMLV)-based retroviral vector expressing the murine (1,3)GT gene. Endpoints of the study include safety assessments, efficacy, and immunological responses.

ELIGIBILITY:
Inclusion Criteria:

* Histological/cytological diagnosis of melanoma. AJCC stage IV (any T, any N, M1), metastatic, progressive, refractory, melanoma.
* Patients may have advanced unresectable stage IV disease, resectable stave IV disease or recently resected stage IV disease (<10 weeks prior) with no apparent disease.
* Eastern Cooperative Oncology Group (ECOG) Performance Status ≤1.
* Serum albumin ≥3.0 gm/dL.
* Adequate organ function including:

  * A. Marrow: Hemoglobin ≥10.0 gm/dL, absolute granulocyte count (AGC) ≥1,000/mm3, platelets ≥75,000/mm3, absolute lymphocyte count ≥475/mm3.
  * B. Hepatic: Serum total bilirubin ≤2.5 x upper limit of normal (ULN), ALT (SGPT) and AST (SGOT) ≤2.5 x ULN.
  * C. Renal: Serum creatinine (sCr) ≤ 1.5 x upper limit of normal.
* Prior therapy for melanoma that may include surgery, radiation therapy, immunotherapy including interleukins and interferon, and/or ≤2 different regiments of systemic chemotherapy, targeted therapy, or other experimental systemic therapies. Prior treatment with immune checkpoint inhibitors is not allowed.
* Patients must be ≥4 weeks since major surgery, radiotherapy, chemotherapy (6 weeks if they were treated with nitrosureas) or biotherapy/targeted therapies.
* Patients must have the ability to understand the study, its risks, side effects, potential benefits and be able to give written informed consent to participate. Patients may not be consented by a durable power of attorney (DPA).
* Male and female subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental drug, and for one month after the last immunization.

Exclusion Criteria:

* Age <18-years-old.
* Active CNS metastases or carcinomatous meningitis. Patients with CNS lesions that have been treated and who have no evidence of progression in the brain on CT/MRI for

  ≥1 month are eligible. Pregnant or nursing women due to the unknown effects of immunization on the developing fetus or newborn infant.
* Other malignancy within five years, except the following may be eligible:

  * patients curatively treated for localized squamous or basal cell carcinoma of the skin or for carcinoma in situ of the uterine cervix (CIN) or breast,
  * patients with a history of malignant tumor who have been disease free for at least five years and are not currently being treated.
* History of an allogeneic solid organ transplant or bone marrow transplant, or current active immunosuppressive therapy such as cyclosporine, tacrolimus, etc.
* Subjects taking systemic (parentally or orally) corticosteroid therapy for any reason, including replacement therapy for hypoadrenalism, are not eligible. Topical steroids are acceptable as are intranasal steroids.
* Active infection or antibiotics within 48 hours prior to study enrollment, including unexplained fever (temp > 38.1°C), if deemed clinically significant by the treating physician.
* Evidence of active autoimmune disease (e.g., systemic lupus erythematosis, rheumatoid arthritis, with the exception of vitiligo. Patients with a remote history of asthma or mild asthma are eligible.
* Other serious medical conditions that may be expected to limit life expectancy to less than 2 years (e.g., liver cirrhosis).
* Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc).
* Patients having previously undergone splenectomy.
* Patients with known hepatitis or unstable liver disease, and/or positive serologies for Hepatitis B or C and HIV.
* Patients with sickle-cell anemia or thalassemia major.
* Subjects who received prior treatment with immune checkpoint inhibition, consisting of ipilimumab, tremelimumab, nivolumab, pembrolizumab or other antibody to CTLA4 or PD-1.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2014-06; Primary Completion 2018-04-05 (Actual); Study Completion 2021-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene Kennedy, MD, Study Director — NewLink Genetics Corporation
Locations (5):
- United States (5):
  - Oncology Specialists, Niles, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - University of Kansas Cancer Center, Westwood, Kansas
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Tennessee Medical Center, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The enrollment and treatment phase of this trial was terminated early, but the FDA required 15 year long term follow-up for gene therapy is still ongoing.
Groups:
- Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab: Arm 1A will receive ipilimumab at 3 mg/kg given every 3 weeks for 4 weeks and 300 Million HyperAcute®-Melanoma (HAM) Immunotherapy cells per each immunization, given every week for 4 weeks, every 2 weeks for 5 months, every month for 6 months, and every 3 months for one year.
  HyperAcute®-Melanoma (HAM) Immunotherapy
  Ipilimumab
- Arm 2A Ipilimumab Alone: Arm 2A will receive ipilimumab alone at 3 mg/kg every 3 weeks for a total of four doses.
  Ipilimumab
- Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab: Arm 1B will receive nivolumab alone at 3 mg/kg given every 2 weeks and 300 Million HyperAcute®-Melanoma (HAM) Immunotherapy cells per each immunization, given every week for 4 weeks, every 2 weeks for 5 months, every month for 6 months, and every 3 months for one year.
  HyperAcute®-Melanoma (HAM) Immunotherapy
  Nivolumab
- Arm 2B Nivolumab Alone: Arm 2B will receive nivolumab alone at 3 mg/kg given every 2 weeks
  Nivolumab
- Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab: Arm 1C will receive pembrolizumab at 2 mg/kg given every 3 weeks and 300 Million HyperAcute®-Melanoma (HAM) Immunotherapy cells per each immunization, given every week for 4 weeks, every 2 weeks for 5 months, every month for 6 months, and every 3 months for one year.
  HyperAcute®-Melanoma (HAM) Immunotherapy
  Pembrolizumab
- Arm 2C Pembrolizumab Alone: Arm 2C will receive pembrolizumab at 2 mg/kg given every 3 weeks
  Pembrolizumab
Period: Overall Study
Arm/Group | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab | Arm 2A Ipilimumab Alone | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab | Arm 2B Nivolumab Alone | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab | Arm 2C Pembrolizumab Alone
Started | 11 | 16 | 6 | 6 | 5 | 3
Completed | 2 | 11 | 0 | 0 | 0 | 0
Not Completed | 9 | 5 | 6 | 6 | 5 | 3
Not completed — Adverse Event | 1 | 4 | 2 | 1 | 1 | 0
Not completed — Lack of Efficacy | 7 | 0 | 2 | 1 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 2 | 1 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 1
Not completed — Study terminated by Sponsor | 0 | 0 | 2 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab | Arm 2A Ipilimumab Alone | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab | Arm 2B Nivolumab Alone | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab | Arm 2C Pembrolizumab Alone | Total
Number analyzed (Participants) | 11 | 16 | 6 | 6 | 5 | 3 | 47
Age, Continuous [Mean (Full Range); unit: years] | 59.5 [39 to 75] | 63.4 [49 to 86] | 61.3 [37 to 80] | 67.5 [57 to 75] | 60.8 [53 to 77] | 62.3 [56 to 72] | 62.4 [37 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 3 | 2 | 3 | 1 | 17
  Male | 7 | 12 | 3 | 4 | 2 | 2 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 11 | 16 | 6 | 6 | 5 | 3 | 47
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 11 | 16 | 6 | 6 | 5 | 3 | 47
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
ECOG Performance Status [Count of Participants; unit: Participants] — GRADE ECOG PERFORMANCE STATUS
  0 - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. - Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. - Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. - Dead
  Participants
    ECOG PS Score 0 | 10 | 10 | 4 | 3 | 4 | 2 | 33
    ECOG PS Score 1 | 1 | 6 | 2 | 3 | 1 | 1 | 14

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability Assessed by Development of AEs and Laboratory Parameters
Description: To determine the safety of administration of immune checkpoint inhibition consisting of ipilimumab, nivolumab, or pembrolizumab with or without dorgenmeltucel-L immunotherapy for patients with stage IV melanoma
Time Frame: 2 years
Population: The primary population for safety analyses is the safety analysis set, defined as all randomized subjects who receive at least one administration of study treatment (dorgenmeltucel-L or immune checkpoint therapy).
Measure: Number; unit: participants with event
Arm/Group | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab | Arm 2A Ipilimumab Alone | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab | Arm 2B Nivolumab Alone | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab | Arm 2C Pembrolizumab Alone
Number analyzed (Participants) | 11 | 16 | 6 | 6 | 5 | 3
participants with event
  At least one TEAE | 11 | 16 | 6 | 5 | 5 | 3
  At least one Serious TEAE | 3 | 3 | 1 | 2 | 0 | 2
  At least one DLT | 0 | 0 | 0 | 0 | 0 | 0
  At least one severe TEAE | 7 | 6 | 4 | 2 | 1 | 1
  At least one related TEAE | 11 | 0 | 6 | 0 | 5 | 0
  At least one TEAE leading to discontinuation | 1 | 4 | 2 | 1 | 1 | 0

2. Primary Outcome: Clinical Response Rate
Description: To estimate the clinical response rate of metastatic melanoma patients after immunotherapy with dorgenmeltucel-L immunotherapy plus immune checkpoint inhibition
Time Frame: 2 years
Population: The enrollment and treatment phase of this trial was terminated early. The analysis of clinical response rate was limited as enrollment to the trial was closed early.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab | Arm 2A Ipilimumab Alone | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab | Arm 2B Nivolumab Alone | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab | Arm 2C Pembrolizumab Alone
Number analyzed (Participants) | 8 | 14 | 4 | 2 | 4 | 3
Participants | 2 | 4 | 1 | 0 | 2 | 1

ADVERSE EVENTS:
Time Frame: All AEs were collected occurring during the study period from the time of the first dose to the last day of the 30-day post-treatment follow-up period.
Arm/Group | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab | Arm 2A Ipilimumab Alone | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab | Arm 2B Nivolumab Alone | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab | Arm 2C Pembrolizumab Alone
All-Cause Mortality (participants affected / at risk) | 5/11 | 7/16 | 2/6 | 1/6 | 1/5 | 2/3
Serious Adverse Events (participants affected / at risk) | 3/11 | 3/16 | 1/6 | 2/6 | 0/5 | 2/3
Other Adverse Events (participants affected / at risk) | 11/11 | 16/16 | 6/6 | 5/6 | 5/5 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab (N=11) | Arm 2A Ipilimumab Alone (N=16) | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab (N=6) | Arm 2B Nivolumab Alone (N=6) | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab (N=5) | Arm 2C Pembrolizumab Alone (N=3)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gallbladder pain (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1A HyperAcute®-Melanoma (HAM) + Ipilimumab (N=11) | Arm 2A Ipilimumab Alone (N=16) | Arm 1B HyperAcute®-Melanoma (HAM) + Nivolumab (N=6) | Arm 2B Nivolumab Alone (N=6) | Arm 1C HyperAcute®-Melanoma (HAM) + Pembrolizumab (N=5) | Arm 2C Pembrolizumab Alone (N=3)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0 | 2 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Angina Pectoris (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Myocarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 2 | 1 | 1 | 0 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0
Ear Haemorrhage (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Middle Ear Inflammation (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypophysitis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 1 | 1 | 0 | 0
Eye Discharge (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Watering Eyes (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal distention (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Abdominal Pain (Gastrointestinal disorders) | 0 | 2 | 2 | 1 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 3 | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Gastoesophaeal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0 | 0
Gingival Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0
Lip pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Melaena (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 9 | 3 | 4 | 4 | 2 | 0
Oral Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Stomach Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1 | 5 | 3 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 2 | 0 | 2 | 0 | 0 | 0
Chills (General disorders) | 5 | 1 | 1 | 0 | 1 | 0
Fatigue (General disorders) | 9 | 7 | 5 | 3 | 5 | 2
Inflammation (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Injection site erythema (General disorders) | 11 | 0 | 6 | 0 | 4 | 0
Injection site induration (General disorders) | 9 | 0 | 4 | 0 | 5 | 0
Injection site irritation (General disorders) | 4 | 0 | 2 | 0 | 4 | 0
Injection site pain (General disorders) | 9 | 0 | 5 | 0 | 0 | 0
Injection site Pruritus (General disorders) | 8 | 0 | 6 | 0 | 2 | 0
Injection Site Reaction (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 11 | 0 | 5 | 0 | 4 | 0
Injection site warmth (General disorders) | 6 | 0 | 4 | 0 | 1 | 0
Malaise (General disorders) | 3 | 0 | 1 | 1 | 0 | 1
Mucosal Inflammation (General disorders) | 1 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 1 | 1 | 2 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 4 | 3 | 2 | 2 | 1 | 0
Gallbladder pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 1
Autoimmune disorder (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hypersensitivity (Immune system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ear Infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 0 | 0 | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0 | 0 | 0
Incision Site Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2 | 0 | 1 | 1 | 1
Aspartate Aminostransferase Increased (Investigations) | 0 | 1 | 0 | 2 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 3 | 1 | 1 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 4 | 1 | 0 | 0
Blood immunoglobulin E increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood immunoglobulin G increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone decreased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 2 | 0 | 0 | 1 | 0
Cortisol increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein Increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 0 | 1 | 0
Thyroxine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Weight Decreased (Investigations) | 1 | 1 | 1 | 0 | 0 | 0
Weight Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 2 | 3 | 1 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 1 | 2 | 1 | 0 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 3 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0 | 1 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 2 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0
bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2 | 0 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 0 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Neck Mass (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 3 | 0 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 1
Cognitive Disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 5 | 4 | 3 | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 4 | 4 | 5 | 2 | 2 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
IIIrd nerve disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Tinnitus (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
agitation (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 1 | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 4 | 1 | 1 | 1 | 0
Libido decreased (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Acute Kidney Injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Polyuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Breast Discharge (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 | 0 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1 | 2 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 2 | 2 | 0
dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 1 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Maculopapular Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 2 | 1 | 0 | 0
Night Sweats (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 10 | 4 | 2 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 4 | 2 | 1 | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Skin Mass (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0
Yellow Skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. The enrollment and treatment phase of this trial was terminated early and the IND has been closed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT02054520/Prot_SAP_000.pdf